CLINICAL TRIAL: NCT07175337
Title: Effect of Maryam Plant and Surah on Birth Pain, Anxiety and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Esra Sayar, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AtaturkU-SBF-ES-02
Record Dates: First submitted 2025-08-21; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy; No Pregnancy Complications; Cervical Dilatation of 4-6 cm (Early Active Phase); Muslim
Keywords: Virgin Mary's Hand Plant; Surah Maryam; Labor Pain; Birth Anxiety; Birth Satisfaction
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The research was conducted in a randomized controlled experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surah Maryam group (Experimental): Pregnants who came for birth were taught the Surah Maryam. They were monitored throughout the labor process, and in addition to routine midwifery care, the Surah Maryam was recited twice during labor to provide spiritual support.
  Interventions: Behavioral: Surah Maryam group
- Virgin Mary's Hand Plant group (Experimental): By monitoring the labor throughout the process, in addition to routine midwifery care, the pregnant was provided with moral support by placing the Virgin Mary's Hand plant in water and watching the plant unfold, guiding her to the idea that the birth canal would also open in the same way.
  Interventions: Behavioral: Virgin Mary's Hand Plant Group
- Control Group (No Intervention): Routine midwifery care was provided at birth

INTERVENTIONS:
Behavioral: Surah Maryam group — Pregnant women who came for birth were taught Surah Maryam. They were monitored throughout the labor process, and in addition to routine midwifery care, Surah Maryam was played twice during labor to provide spiritual support.
  Arms: Surah Maryam group
Behavioral: Virgin Mary's Hand Plant Group — he pregnant woman was monitored throughout labor; in addition to routine midwifery care, she was given spiritual support by placing the Virgin Mary's Hand plant in water and watching the plant unfold, encouraging her to believe that the birth canal also opens in the same way.
  Arms: Virgin Mary's Hand Plant group

SUMMARY:
This randomized controlled trial was conducted to determine the effects of spiritual support provided by Virgin Mary's hand plant and Surah Maryam on labor anxiety, labor pain, and satisfaction.

DETAILED DESCRIPTION:
No other study has been found investigating the effects of both the Maryam Surah and the Virgin Mary plant on labor anxiety, labor pain, and labor satisfaction. The effects of the parameters to be examined in this project have not yet been examined, and the effects of the Maryam Surah recited to pregnant women during labor and the Virgin Mary plant, believed to help open the birth canal, have not been tested. The study aims to contribute to the literature through a randomized controlled trial and to obtain data that will inform future studies.

ELIGIBILITY:
Inclusion Criteria:

* • Being literate

  * Being open to communication
  * Being at term (37-40 weeks)
  * Having a single, live fetus
  * Having no pregnancy complications
  * Having no conditions preventing labor
  * Having 4-6 cm cervical dilation (early active phase)
  * Planning a vaginal birth
  * Not having a diagnosed psychiatric illness
  * Volunteering to participate in the study
  * Being in cephalic presentation
  * Being Muslim

Exclusion Criteria:

* Being illiterate

  * Having a high-risk pregnancy
  * Having a planned cesarean section
  * Developing complications during labor
  * Using pain-reducing methods such as narcotic analgesics or sedatives
  * Having a diagnosed psychiatric illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Enrollment: 125 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | through study completion, an average of 1 year
  VAS is used to measure perceived pain. It consists of a 10 cm (100 mm) line with one end labeled "no pain" and the other "worst possible pain." The participant marks a point on the line corresponding to the intensity of their pain. The distance in millimeters from "no pain" to the mark is measured and recorded as the pain score. Cline et al. (1992) reported that vertical orientation was better understood by patients. The scale was originally developed by Price et al. (1983). Eti-Aslan (1998) found that VAS was more sensitive in the evaluation of postoperative (acute) pain
Oxford Worry About Labour Scale (OWLS) | Through study completion, an average of 1 year
  Developed by Redshaw, Martin, Rowe, and Hockley (2009) to assess women's worries related to the childbirth process. The Turkish validity and reliability study was conducted by Erkal and Özentürk (2016). The scale consists of 10 items rated on a 4-point Likert scale: (1) Very worried, (2) Fairly worried, (3) Not very worried, (4) Not at all worried. Scores are calculated from the total (minimum = 10, maximum = 40). The scale has three subdimensions: Pain and Distress, Uncertainty Before Birth, and Interventions. The Cronbach's alpha reliability coefficient of the Turkish version was found to be 0.83 (Erkal Aksoy & Özentürk, 2016). In this study, the Cronbach's alpha value of the questionnaire was found to be 0.75.
Birth Satisfaction Scale-Revised (BSS-R) | through study completion, an average of 1 year
  The original Birth Satisfaction Scale was developed by Martin and Fleming (2011) to assess women's satisfaction with childbirth. In 2013, Martin and Martin revised the scale by reducing the number of items, resulting in the Birth Satisfaction Scale-Revised (BSS-R). The BSS-R is a 10-item Likert-type scale rated as: Strongly agree (4 points), Agree (3 points), Neutral (2 points), Disagree (1 point), Strongly disagree (0 points). Items 2, 4, 7, and 8 are reverse-scored. The total score ranges from 0 to 40, with higher scores indicating greater satisfaction. The scale has three subdimensions: Quality of Care (communication, support from healthcare providers, and cleanliness of the delivery room), Women's Personal Attributes (sense of control and anxiety during childbirth), and Stress Experienced During Labor (perceived stress and duration of labor). The Cronbach's alpha reliability coefficient of the Turkish version was reported as 0.72 (Gökmen, 2017). In this study, the Cronbach's alpha

CONTACTS AND LOCATIONS:
Overall Officials: WHO, Study Director — World Health Organization; ICMJE ICMJE, Study Director — ICMJE
Locations (1):
- Ataturk Universty, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results of this study will be made available upon reasonable request. Data will be shared beginning , 6 months after publication and ending 5 years following article publication. Access will be granted to researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by the study investigators. Data will be shared through \[specify repository or method of sharing].
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available beginning 6 months after publication and ending 5 years] following publication.
Access Criteria: Access to de-identified individual participant data will be granted to researchers with a methodologically sound proposal. Requests must include a clear research question and analysis plan. Approval will be required from the study's principal investigator before data are released.
URL: https://outlook.live.com/mail/0/id/AAkALgAAAAAAHYQDEapmEc2byACqAC%2FEWg0AkmF%2FszhosUe9os%2FLB9EsbAAI8XaE8gAA